CLINICAL TRIAL: NCT07242690
Title: Advancing PET-CT Imaging With Photon Counting Detector CT
Brief Title: PET-CT Imaging With PCD-CT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team is working on contracts.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Kevin Horn, Research Instructor-Faculty, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: Pro00146888
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer (H&N)
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PET CT scan (Other): To compare the image quality of PET images constructed using non-contrast PCD-CT image data to PET images constructed using conventional standard-of-care non-contrast EID-CT image data by performing a quantitative analysis of measurable image quality parameters.
  Interventions: Other: PCD-CT
- PCD-CT (Other): To compare the subjective image quality of PET images constructed using non-contrast PCD-CT image data to PET images constructed using conventional standard-of-care non-contrast EID-CT image data by performing a qualitative analysis of diagnostic confidence as determined by board-certified radiologists/nuclear medicine physicians during image review.
  Interventions: Other: PET CT

INTERVENTIONS:
Other: PCD-CT — A direct qualitative comparison of the subjective PET image quality will be performed.
  Two blinded board-certified radiologists/nuclear medicine physicians will independently review PET images constructed using non-contrast PCD-CT data as well as PET images constructed using standard of care non-contrast EID-CT data in random order. Both raters will assess PET images subjectively regarding overall image quality using a five-point Likert scale. The rating will be defined as: (1) non-diagnostic - insufficient diagnostic confidence, (2) poor - low diagnostic confidence, (3) moderate - average diagnostic confidence; (4) good - high diagnostic confidence, and (5) excellent - full diagnostic confidence.
  Arms: PET CT scan
Other: PET CT — To compare the subjective image quality of PET images constructed using non-contrast PCD-CT image data to PET images constructed using conventional standard-of-care non-contrast EID-CT image data by performing a qualitative analysis of diagnostic confidence as determined by board-certified radiologists/nuclear medicine physicians during image review.
  Arms: PCD-CT

SUMMARY:
This pilot study evaluates the clinical utility of photon counting detector computed tomography (PCD-CT) in PET-CT imaging for head and neck cancer. Twenty adult patients undergoing standard-of-care PET-CT will also receive PCD-CT imaging. The study compares image quality and diagnostic confidence between conventional energy-integrating detector CT (EID-CT) and PCD-CT for attenuation correction and anatomical imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for or completed standard-of-care PET-CT of head and neck within ≤30 days

Exclusion Criteria:

* Non-diagnostic PET-CT
* Intervening therapy between scans
* Iodinated contrast allergy
* Renal insufficiency (GFR < 45)
* Pregnancy
* Gross motion artifacts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
improve PET image w/ non-contrast PCD-CT data | 2 years
  We expect that the subjective PET image quality will be improved by using non-contrast PCD-CT data for construction resulting in higher diagnostic confidence; demonstrating a case for the integration of PCD-CT into standard of care clinical PET-CT imaging in the future. There will be no direct benefit to study participants and the outcome will not be directly reported to the treatment team or patient and will not impact treatment or care received.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Horn, PhD, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States